CLINICAL TRIAL: NCT04536441
Title: Effects of an Ultra-brief Online Mindfulness-based Intervention on Mental Health During the Coronavirus Disease (COVID-19) Outbreak in Malaysia: A Randomised Controlled Trial
Brief Title: Ultra-brief Online Mindfulness-based Intervention During COVID-19 Movement Control Order
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Collaborators: Sunway University (Other)
Responsible Party: Principal Investigator, Pheh Kai Shuen, Lecturer, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U/SERC/62/2020
Record Dates: First submitted 2020-08-26; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Mental Health Wellness; Psychological Security; Psychological Distress
Keywords: Mindfulness; Online Intervention; COVID-19; Movement Control Order
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Ultra Brief Online Mindfulness-based Intervention
  Interventions: Behavioral: Ultra Brief Online Mindfulness-based Intervention
- Control (Placebo Comparator): This arm requires participants to answer questions about themselves.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Ultra Brief Online Mindfulness-based Intervention — We adapted and contextualized the original RAIN protocol to local pandemic-induced lockdown situation, with short journaling prompts that engage participants in self-reflection. Journaling is known to be a creative way to engage people in a therapeutic activity which promotes self-awareness (Utley & Garza, 2011). Creating a visual narration of thoughts, feelings and experiences help individuals make internal experiences more tangible and manageable, especially during these uncertain times.
  Arms: Treatment
Behavioral: Control — The control group participants were asked to report preventive measures that they have taken to prevent COVID-19, ways that they obtained Movement Control Order news, and things that they wished to do once the Movement Control Order is lifted.
  Arms: Control

SUMMARY:
The federal government of Malaysia implemented a nationwide Movement Control Order (MCO) to control the COVID-19 outbreak. The MCO, however, has been found to have a negative impact on people's mental wellbeing. Interventions that can improve mental health under restricted movement condition is urgently. The present study investigated the impact of a brief, online mindfulness-based intervention on mental health using two-arm randomized controlled trial design. A total of 161 participants self-reported their feeling, anxiety, psychological insecurity, and well-being at baseline (T1) and post-test (T2), while 61 of them answered the same set of measures and the fear of COVID-19 scale in a follow-up study two weeks later (T3).

ELIGIBILITY:
Inclusion Criteria:

* People residing in Malaysia during the Movement Control Order.

Exclusion Criteria:

* People who are unable to read or write in either Malay, English or Mandarin languages.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes of Subjective Unit of Distress | It was measured at pre-intervention, post-intervention (through intervention completion, on average 10 minutes), and 2-week follow up.
  This is being measured with the Subject Unit of Distress Scale.
Changes of Anxiety Scores | It was being It was measured at pre-intervention, post-intervention (through intervention completion, on average 10 minutes), and 2-week follow up.
  This is being measured with the GAD-7 questionnaire.
Changes of Psychological Insecurity | It was being It was measured at pre-intervention, post-intervention (through intervention completion, on average 10 minutes), and 2-week follow up.
  This is being measured with the Psychological Insecurity Scale.

SECONDARY OUTCOMES:
Changes of General Well-being | It was being It was measured at pre-intervention, post-intervention (through intervention completion, on average 10 minutes), and 2-week follow up.
  This is being measured with the WHO-5 Well-being Index questionnaire.
Fear of COVID-19 | It was being measured at 2-week follow up.
  This is being measured with the Fear of COVID-19 Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Shuen Pheh, MClinPsych, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Universiti Tunku Abdul Rahman, Kampar, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be become available once the study is being published, for 5 years.
Access Criteria: The data will be made available upon request to the corresponding author.